CLINICAL TRIAL: NCT00815568
Title: Prospective Phase II Clinical Trial of Myeloablative Conditioning Regimen With Fludarabine and Busulfan Plus 400 cGy Total Body Irradiation for Hematologic Malignancies
Brief Title: Feasibility and Efficacy Study of Conditioning Regimen for Allogeneic Hematopoietic Cell Transplantation (HCT) With Fludarabine, Busulfan, and Total Body Irradiation (TBI)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Dong Hwan Kim, Dept of Hematology/Medical Oncology, Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-07-020
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Last update posted 2008-12-30 (Estimated); Status verified 2008-12

CONDITIONS: AML; MDS; ALL; CML; Lymphoma
Keywords: fludarabine; busulfan; total body irradiation; conditioning regimen
MeSH Terms: conditions — Lymphoma | interventions — fludarabine phosphate; Busulfan; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regimen (Experimental): Conditioning regimen for AML with FLT3 mutation, AML/MDS unfavorable cytogenetic risk group, chemorefractory NHL or HD, or ALL/CML
  Interventions: Drug: fludarabine phosphate, busulfan

INTERVENTIONS:
Drug: fludarabine phosphate, busulfan — Fludarabine ( 30mg/m2, iv, D-7~D-2) Busulfan (3.2mg/kg, iv, D-6~D-3) Total body irradiation (200cGy/day, D-2,-1)
  Other Names: Fludarabine (Fludara®, Berlex Laboratories, Richmond, CA)

SUMMARY:
The purpose of this study is to evaluate the OS, RFS, and TRM after HCT with low-dose total body irradiation, fludarabine, and busulfan conditioning.

DETAILED DESCRIPTION:
Conventional allogeneic hematopoietic cell transplantation (HCT) for patients with hematological malignancies involves conditioning with high doses of systemic chemo/radiation therapy such as cyclophosphamide (CY) plus 1200 or 1000 cGy total body irradiation (TBI; CY/TBI) or busulfan (Bu) / CY (BuCy). Unfortunately, such regimens have been associated with significant toxicities, limiting their use to otherwise healthy, relatively young patients.

Recently, Fludarabine plus 4 day dose of busulfan (FluBu4) containing myeloablative regimen has been introduced successfully without increasing transplant-related mortality (TRM). To improve transplant outcomes without increasing the risk of recurrence, Russell et al introduced 400cGy of TBI with antithymocyte (ATG, 4.5mg/Kg) into FluBu4 regimen with successful outcomes.

ELIGIBILITY:
Inclusion Criteria:

* At least 15 years old and not more than 65 years old.
* ECOG performance status 0-2.
* Patients with AML or MDS with intermediate/unfavorable cytogenetics.
* Patients with ALL and CML ineligible for Cy/TBI conditioning.
* Patients with NHL or HD eligible to myeloablative HCT.
* Patients receiving unrelated BMT for AML, MDS, ALL, CML, NHL or HD.
* Consent form signed and dated prior to study specific procedures.
* Subject able to comply with the scheduled follow-up and with the management of toxicities.

Exclusion Criteria:

-

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2008-08; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
progression free survival | one year

SECONDARY OUTCOMES:
relapse of primary disease, overall survival, and occurrence of acute/chronic GVHD | one year

CONTACTS AND LOCATIONS:
Overall Officials: Dong Hwan Kim, Study Director — Samsung Medical Center
Locations (1):
- Dong Hwan Kim, Seoul, South Korea